CLINICAL TRIAL: NCT06755619
Title: CtDNA for Early Response Assessment in PCNSL Treated with 1st Line Curative Intent (NLG-PCNSL-01)
Acronym: CAPCI
Status: Recruiting | Type: Observational
Sponsor: Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: 24020; NLG-PCNSL-01 (Other: Tampere University Hospital)
Record Dates: First submitted 2024-12-04; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Primary Central Nervous System (CNS) Lymphoma
Keywords: PCNSL; ctDNA
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Spinal fluid, peripheral blood, tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an international, prospective, multicenter trial with the aim of characterizing circulating tumor DNA (ctDNA) for early response assessment in PCNSL patients treated with standard of care (SOC) 1st line therapy with a curative intent (Figure 1). Secondary endpoints are to assess the clinical characteristics, health-related quality of life (HRQoL), neurological status, and outcome of newly diagnosed primary central nervous system lymphoma (PCNSL) patients in the Nordic countries. Patients eligible for a curative intent SOC 1st line therapy, such as MATRix + high-dose chemotherapy and autologous stem cell transplantation (HDCT/ASCT), are eligible for the trial. Diagnostic tumor tissue, cerebrospinal fluid (CSF), and plasma samples are collected for ctDNA and translational analyses with the aim describing new prognostic and predictive biomarkers. Treatment responses are assessed with the International PCNSL Collaborative Group (IPCG) response criteria, and diagnostic and response assessment magnetic resonance imaging (MRI) images are centrally analyzed in order to describe new prognostic and predictive markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years at diagnosis
* Histologically or cytologically verified diffuse large B-cell lymphoma (DLBCL) of the central nervous system (CNS)
* No prior treatment for PCNSL (pre-treatment corticosteroids are allowed and recommended)
* Fit for standard of care (SOC) 1st line therapy with a curative intent such as full-dose MATRix, according to local policy
* Able to give voluntary written informed consent
* If the patient is temporarily incapacitated to give the voluntary written informed consent, due to PCNSL, the informed consent can be obtained from a legally acceptable representative, according to the International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use - Guideline for Good Clinical Practice (ICH-GCP) guidelines

Exclusion Criteria:

* Lymphoma outside the CNS
* History of prior hematological malignancy e.g. low grade B-cell lymphoma
* Psychiatric illness or condition, other than PCNSL, which could interfere with the ability to understand the requirements of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed primary central nervous system diffuse large B-cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA | 6 months from initiation of 1st line therapy
  Predictive value and sensitivity of CSF and plasma ctDNA

CONTACTS AND LOCATIONS:
Locations (5):
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Undecided